CLINICAL TRIAL: NCT02159573
Title: A Multicenter, Retrospective, Observational Study Evaluating Real-world Clinical Outcomes in Relapsing-remitting Multiple Sclerosis Patients Who Transition From Tysabri® (Natalizumab) to Tecfidera® (Dimethyl Fumarate)
Brief Title: Real-world Outcomes on Tecfidera (BG00012, Dimethyl Fumarate) Post-Tysabri (BG00002, Natalizumab)
Acronym: STRATEGY
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: 109MS412; US-BGT-13-10564 (Other: BIIB GMA)
Record Dates: First submitted 2014-05-19; First posted 2014-06-10 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2016-06

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Natalizumab; Dimethyl Fumarate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: natalizumab — Administered as per routine clinical practice
  Other Names: BG00002; Tysabri
Drug: dimethyl fumarate — Administered as per routine clinical practice
  Other Names: BG00012; Tecfidera; DMF

SUMMARY:
The primary objective of the study is to evaluate relapse activity, as measured by the proportion of participants relapsed at 12 months, in participants with relapsing-remitting multiple sclerosis (RRMS) who transition from Tysabri (BG00002) to Tecfidera (BG00012) in the real-world setting. The secondary objective is to further evaluate relapse activity, defined as annualized relapse rate (ARR), hospitalization and intravenous corticosteroid use, during the first year of Tecfidera treatment following transition from Tysabri treatment.

DETAILED DESCRIPTION:
The study period will consist of a single time point retrospective medical chart abstraction with no required study visits or procedures. Data collection for this study is expected to last up to approximately five months.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of RRMS per McDonald criteria
* Received at least 12 months of continuous treatment with Tysabri monotherapy prior to initiation of Tecfidera. Note: continuous treatment with Tysabri is defined as treatment uninterrupted by other disease-modifying treatment.
* Initiated treatment with Tecfidera at least 12 months prior to enrollment into the study
* Patient has sufficient available medical records for data abstraction to meet the objectives of the study

Key Exclusion Criteria:

* Diagnosed with a progressive form of multiple sclerosis (MS) (progressive-relapsing, primary progressive, secondary progressive)
* Received treatment with any of the following after discontinuation of Tysabri and before initiation of treatment with Tecfidera (i.e., during washout period): interferon-beta, glatiramer acetate, fingolimod, teriflunomide, rituximab, alemtuzumab, ocrelizumab or any investigational compound for the treatment of RRMS
* Received BG00012, or other formulations of dimethyl fumarate, or Fumaderm® or compounded fumarates at any time prior to initiation of treatment with Tecfidera
* History of progressive multifocal leukoencephalopathy (PML) while on Tysabri or within 6 months of discontinuing treatment with Tysabri

NOTE: Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with a diagnosis of RRMS receiving at least 12 months of continuous treatment with Tysabri monotherapy prior to initiation of Tecfidera. Additionally, participants must have initiated treatment with Tecfidera at least 12 months prior to enrollment into the study.
Sampling Method: Non-Probability Sample
Enrollment: 530 (Actual)
Dates: Start 2014-07; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Kaplan-Meier Estimates for the Proportion of Participants relapsed at 12 months after initiation of treatment with Tecfidera | 12 months post initiation of treatment with Tecfidera

SECONDARY OUTCOMES:
ARR at 12 months post-initiation of treatment with Tecfidera | 12 months post initiation of treatment with Tecfidera
The percent of participants with MS-related hospitalization at 12 months post-initiation of treatment with Tecfidera | 12 months post initiation of treatment with Tecfidera
The percent of participants with relapses requiring treatment with intravenous steroids | 12 months post initiation of treatment with Tecfidera

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (43):
- United States (43):
  - Research Site, Birmingham, Alabama
  - Research Site, Cullman, Alabama
  - Research Site, Gilbert, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Aurora, Colorado
  - Research Site, Centennial, Colorado
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Jacksonville Beach, Florida
  - Research Site, Palm Bay, Florida
  - Research Site, Tampa, Florida
  - Research Site, Athens, Georgia
  - Research Site, Atlanta, Georgia
  - Research Site, Idaho Falls, Idaho
  - Research Site, Chicago, Illinois
  - Research Site, Peoria, Illinois
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Glen Burnie, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Farmington Hills, Michigan
  - Research Site, Golden Valley, Minnesota
  - Research Site, Lincoln, Nebraska
  - Research Site, Teaneck, New Jersey
  - Research Site, Amherst, New York
  - Research Site, East Meadow, New York
  - Research Site, New York, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Columbus, Ohio
  - Research Site, Gahanna, Ohio
  - Research Site, Uniontown, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Portland, Oregon
  - Research Site, Altoona, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Nashville, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Newport News, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Seattle, Washington
  - Research Site, Spokane, Washington
  - Research Site, Madison, Wisconsin
  - Research Site, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Cohan SL, Moses H, Calkwood J, Tornatore C, LaGanke C, Smoot KE, Meka V, Okwuokenye M, Hotermans C, Mendoza JP, Mann MK, Meltzer LA. Clinical outcomes in patients with relapsing-remitting multiple sclerosis who switch from natalizumab to delayed-release dimethyl fumarate: A multicenter retrospective observational study (STRATEGY). Mult Scler Relat Disord. 2018 May;22:27-34. doi: 10.1016/j.msard.2018.02.028. Epub 2018 Feb 26. PMID 29524759